CLINICAL TRIAL: NCT00372983
Title: A Randomized, Placebo Controlled, Phase 1b Trial to Evaluate the Safety and Pharmacokinetics of NOV-205 in Chronic Viral Hepatitis C Subjects (Genotype 1) Who Have Failed Treatment With Pegylated Interferon Plus Ribavirin
Brief Title: Safety and PK Study of NOV-205 to Treat Chronic HCV Who Fail Standard Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cellectar Biosciences, Inc. (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NOV205-C101
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Hepatitis C
Keywords: chronic HCV; Failed treatment; genotype 1; failed treatment with pegylated interferon plus ribavirin
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: NOV-205

SUMMARY:
The purpose of this research trial is to find out whether NOV-205 is well tolerated compared to placebo (salt water) in people with hepatitis C. In addition, this trial will test how NOV-205 is absorbed by your body after single and multiple doses of the trial drug, and it will look for early signs of therapeutic activity (decreases in indicators in the blood for the hepatitis C virus and for liver damage). This is known as pharmacokinetics (PK). NOV-205 is an experimental drug. "Experimental" means that the trial drug is currently being tested and is not approved for sale in the United States by the Food and Drug Administration (FDA). However, NOV-205 has been approved by the Russian Federation for treatment of liver diseases including hepatitis C. Clinical studies in that country showed that subjects treated with NOV-205 alone had decreased indicators in the blood for the hepatitis C virus and for liver damage.

DETAILED DESCRIPTION:
This Phase 1b trial aims to evaluate the pharmacokinetic profile of NOV-205, and in comparison to placebo, identify early signs of antiviral activity (with a quantitative reduction of >0.5 log10 in serum HCV RNA level (Elbeik, 2004)) and establish a safety profile of NOV-205 as monotherapy in subjects with chronic HCV who are non-responders to treatment with pegylated interferon plus ribavirin. This trial will also explore the effect of NOV-205 on serum biochemical markers of liver damage (e.g. alanine aminotransferase, ALT) as indications of biologic activity. Results of this trial will guide the design of future Phase 2 studies of NOV-205 in chronic hepatitis C subjects.

ELIGIBILITY:
Inclusion Criteria:

* A serum HCV RNA level of >100,000 IU/ml using a quantitative, branched-chain-DNA (bDNA)-based assay (lower limit of quantitation = ~650 IU/ml) or other equally sensitive quantitative methods.
* Infection with genotype 1 HCV
* Documented failure to respond to treatment (defined as a patient who did not achieve an early viral response (EVR) (≥2 log reduction in serum HCV RNA or undetectable HCV RNA after 12 weeks of treatment) OR is serum HCV RNA positive after 24 weeks of treatment with pegylated interferon plus ribavirin for hepatitis C.
* Women of childbearing potential willing to use two acceptable methods of birth control during trial participation or are sterile or post-menopausal (defined as not having a menstrual cycle for greater than two years)
* Sexually active male subjects are practicing acceptable methods of contraception during trial participation
* Have the ability to understand the requirements of the trial, have provided written informed consent, and agree to abide by the trial restrictions and to return for the required assessments
* The subject must be able to self administer daily subcutaneous injections or their caregiver must be able to administer daily subcutaneous injections

Exclusion Criteria:

* Clinical, laboratory, or histological evidence of liver cirrhosis
* Evidence of hepatic decompensation (presence of or a history of ascites, hepatic encephalopathy, variceal bleeding, or hepatocellular carcinoma)
* Co-infection with human immunodeficiency virus (HIV) or active hepatitis B virus (HBV) (as determined by presence of hepatitis B surface antigen (HBsAg)
* Have received pegylated interferon and/or ribavirin within the 60 days prior to randomization
* Any known preexisting medical condition that could interfere with the subject's participation in and completion of the protocol
* Pregnant female or nursing mother

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-08; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetic profile of different dosing regimens of NOV-205.
To establish the safety profile of NOV-205 in comparison to that of placebo.
To compare changes in viral load after treatment with NOV-205 or placebo (as evidenced by a quantitative reduction of >0.5 log10 in serum HCV RNA levels by quantitative analysis as compared to the average of the screening and baseline values).
To evaluate the impact of NOV-205 on serum ALT and AST levels in comparison to that of placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Koff, MD, Principal Investigator — University of Massachusetts, Worcester